CLINICAL TRIAL: NCT01512407
Title: Randomised Controlled Trial on Adjuvant Transarterial Chemoembolisation After Curative Hepatectomy for Hepatocellular Carcinoma
Brief Title: RCT on Adjuvant TACE After Hepatectomy for HCC
Acronym: A-TECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Yue Sun, Dr Cheung Yue Sun, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2011.236-T
Record Dates: First submitted 2012-01-14; First posted 2012-01-19 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Randomised controlled trial; Transarterial chemoembolisation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hepatectomy plus TACE (Experimental): Transarterial chemoembolisation will be performed 4 to 6 weeks after hepatectomy
  Interventions: Procedure: Transarterial chemoembolisation using cisplatin-lipiodol mixture
- Hepatectomy alone (No Intervention)

INTERVENTIONS:
Procedure: Transarterial chemoembolisation using cisplatin-lipiodol mixture — Cisplatin-lipiodol mixture was infused through catheter placed at hepatic artery followed by gelfoam embolisation. This is performed 4 to 6 weeks after surgery
  Arms: Hepatectomy plus TACE

SUMMARY:
We hypothesise that the use of transarterial chemoembolisation (TACE) after liver resection in patients with hepatocellular carcinoma can eradicate residual cancer cells in the liver and thus improve survival. The aim of this study is to compare the survival of patients undergoing liver resection plus post-operative TACE versus liver resection alone.

DETAILED DESCRIPTION:
Liver resection is the mainstay of curative treatment for hepatocellular carcinoma (HCC). However, recurrence is common after surgery and most occurs in the liver. Transarterial chemoembolisation (TACE) is an effective palliative treatment for HCC. It involves the infusion of chemotherapeutic agent admixed with iodised oil followed by embolisation of the hepatic arterial flow using small particles. This procedures allows application of smaller dose of chemotherapy concentrated to the liver and thus is well tolerated with minimal side effects. We conduct a randomised controlled trial evaluating the efficacy of using TACE after hepatectomy in HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* HCC patients received curative hepatectomy with negative resection margin
* Age from 18 to 70
* Child-Pugh class A
* ASA class I to III
* ECOG performance status Grade 0 or 1

Exclusion Criteria:

* Patients receiving concomitant local ablation or previous TACE
* Main portal vein tumour thrombus extraction during hepatectomy
* Tumour arising from caudate lobe
* Presence of extra-hepatic disease
* Very early HCC with solitary tumour and size < 2cm
* Impaired liver function with either clinically detected ascites, hepatic encephalopathy, serum albumin < 25g/L or bilirubin > 50micromol/L
* Renal impairment with creatinine > 200micromol/L
* Severe concurrent medical illness persisting > 6 weeks after hepatectomy
* History of other cancer
* Hepatic artery anomaly making TACE not possible
* Allergy to cisplatin or lipiodol
* Pregnant woman
* Informed consent not available

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
1-year recurrence rate | 1-year after hepatectomy
  The 1-year recurrence rate after hepatectomy in both arms of study were compared

SECONDARY OUTCOMES:
Disease-free survival | 5 years after operation
Overall Survival | 5-year after surgery
Complications of transarterial chemoembolisation | 3-month after transarterial chemoembolisation
Health-related quality of life assessment | 1-year after surgery
  The quality of life assessment was measured by Functional Assessment of Cancer Therapy-General (FACT-G) Questionnaire (Chinese version 3)

CONTACTS AND LOCATIONS:
Overall Officials: Yue Sun Cheung, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China